CLINICAL TRIAL: NCT03351569
Title: Intravenous Immunoglobulin for Unverricht-Lundborg Disease: Single-patient Trial.
Brief Title: Intravenous Immunoglobulin for Unverricht-Lundborg Disease.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale di Mantova (Other)
Responsible Party: Principal Investigator, Alfonso Ciccone, MD, Azienda Socio Sanitaria Territoriale di Mantova
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200200; 2017-002147-15 (EudraCT Number)
Record Dates: First submitted 2017-10-27; First posted 2017-11-24 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Unverricht-Lundborg Disease
Keywords: Unverricht-Lundborg disease; progressive myoclonus epilepsy; pharmacoresistant epilepsy
MeSH Terms: conditions — Unverricht-Lundborg Syndrome; Myoclonic Epilepsies, Progressive | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: sigle patient trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drug and placebo had the same appearance and are wrapped in foil paper before being shown to the patient.
  Outcome evaluation is carried out by personnel not involved in the treatment at a distant site, one month after treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunoglobulin (Experimental): Intravenous immunoglobulin 25 grams (five 100 ml bottles, 5g/100ml), in 3 hours, once a month for one year.
  Interventions: Drug: Intravenous immunoglobulin
- Saline solution (Placebo Comparator): Intravenous saline solution 500 ml (five 100 ml bottles), in 3 hours, once a month for one year.
  Interventions: Drug: Intravenous immunoglobulin

INTERVENTIONS:
Drug: Intravenous immunoglobulin — Intravenous drip.
  Other Names: Venital

SUMMARY:
Single patient randomized double blind trial to assess whether intravenous immunoglobulin can improve the clinical outcome of a case suffering from Unverricht-Lundborg disease.

DETAILED DESCRIPTION:
Single patient randomized double blind trial to assess whether intravenous immunoglobulin can improve the clinical outcome of a case suffering from Unverricht-Lundborg disease (clinical and genetic diagnosis).

The patient was randomized to be treated with intravenous immunoglobulin or placebo 1:1 (crossover) once a month for at least one year.

Main objective: improvement of the action myoclonus. Secondary objectives: Improvement in the overall score and in individual sections of the Unified Myoclonus Rating Scale at one year; patient preferences based on results at the end of the trial.

The first analyst was scheduled at one year from the start of the trial. The program was to discuss the patient's analysis data and to let the patient decide in three possible ways: to continue the trial, to continue treatment with immunoglobulins, to suspend the treatment. Depending on the decision, it was planned to follow the patient throughout the year after the analysis, at least for one year.

ELIGIBILITY:
Inclusion Criteria:

* Malattia di Unverricht-Lundborg (genetic diagnosis)

Exclusion Criteria:

* Contraindications to intravenous immunoglobulin

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of at least 20% of the action myoclonus at one year, measured with section 4 (Action Myoclonus) of the Unified Myoclonus Rating Scale. | monthly for one year
  The range for Action Myoclonus Score is 0 (best) - 160 (worst, , i.e. more severe involuntary movements). Percent change = 100 X (Placebo UMRS4 - Treatment UMRS4) / Placebo UMRS4).

SECONDARY OUTCOMES:
Unified Myoclonus Rating Scale (UMRS) overall score improvement. | monthly for one year
  The total value of the UMRS (range from 0 - best - to 365 - worst) is composed of the sum of 6 sections: (1) Patient Questionnaire (range 0-48), (2) Myoclonus at rest (range 0-108), (3) Stimulus Sensitivity (range 0-17), (4) Myoclonus with Action (range 0-160), (5) Functional Tests (0-28), (6) Global Disability Score (range 0-4).
Patient's preference | one year
  The program was to discuss the patient's analysis data with the patient himself and to let him decide in three possible ways: (1) to continue the trial, (2) to continue treatment with immunoglobulins, (3) to suspend the treatment.The choice number 2 is considered a favorable outcome.

IPD SHARING:
Plan to Share IPD: Yes
We planned to publish the results of this single patient trial.

REFERENCES:
- [Background] Lillie EO, Patay B, Diamant J, Issell B, Topol EJ, Schork NJ. The n-of-1 clinical trial: the ultimate strategy for individualizing medicine? Per Med. 2011 Mar;8(2):161-173. doi: 10.2217/pme.11.7. PMID 21695041
- [Background] Guatelli JC, Gingeras TR, Richman DD. Alternative splice acceptor utilization during human immunodeficiency virus type 1 infection of cultured cells. J Virol. 1990 Sep;64(9):4093-8. doi: 10.1128/JVI.64.9.4093-4098.1990. PMID 2384914